CLINICAL TRIAL: NCT02487901
Title: Randomized Controlled Trial: Comparison of Ultrasonic Osteotome and Conventional Drill Osteotome
Brief Title: Comparison of Ultrasonic Osteotome and Conventional Drill Osteotome
Acronym: SONO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SONO1
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Arthrodesis
Keywords: arthrodesiss; cervical vertebra; laminoplasty
MeSH Terms: conditions — Ankylosis | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: ultrasonic bone osteotome
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic osteotome (Active Comparator): making gutter on the hinge side of lamina with ultrasonic osteotome
  Interventions: Device: ultrasonic osteotome
- Drill (Sham Comparator): making gutter on the hinge side of lamina with conventional drill
  Interventions: Device: drill

INTERVENTIONS:
Device: ultrasonic osteotome — making gutter with ultrasonic osteotome
  Other Names: misonix
  Arms: Ultrasonic osteotome
Device: drill — making gutter with drill
  Other Names: electronic drill
  Arms: Drill

SUMMARY:
Ultrasonic bone osteotome has been utilized in various surgical field, but the use in neurosurgery especially in spine surgery is not widely spread. In the present study, the investigators are going to compare bony fusion rate after cervical laminotomy either with ultrasonic osteotome or conventional drill.

DETAILED DESCRIPTION:
Ultrasonic bone osteotome has been utilized in various surgical field, but the use in neurosurgery especially in spine surgery is not widely spread. The tissue selectivity of ultrasonic osteotomy may enhance operative time and reduce tissue trauma. Moreover, bony fusion rate may be increased because of low thermal injury to the bone. In the present study, we are going to compare bony fusion rate after cervical laminotomy either with ultrasonic osteotome or conventional drill.

ELIGIBILITY:
Inclusion Criteria:

1. cervical myelopathy at 3 or more levels due to spondylosis, congenital stenosis, or OPLL;
2. aged more than 20 years
3. with American Society of Anesthesiology physical status class 1 or 2

Exclusion Criteria:

1) concomitant neurological disease such as cerebral palsy or amyotrophic lateral sclerosis; 2) concurrent cancer or infection; 3) previous cervical spinal surgery; 4) a trauma-associated lesion; 5) inability to be followed up (i.e., foreign patients); 6) refusal to participate in the study

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-02-04 (Actual); Study Completion 2018-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo Y, Jeong S, Lee S, Kim TS, Kim JH, Chung CK, Lee CH, Rhee JM, Kong HJ, Kim CH. Machine-learning-based models for the optimization of post-cervical spinal laminoplasty outpatient follow-up schedules. BMC Med Inform Decis Mak. 2024 Sep 30;24(1):278. doi: 10.1186/s12911-024-02693-y. PMID 39350186
- [Derived] Kim CH, Chung CK, Choi Y, Kuo CC, Lee U, Yang SH, Lee CH, Jung JM, Hwang SH, Kim DH, Yoon JH, Paik S, Lee HJ, Jung S, Park SB, Kim KT, Park HP. The Efficacy of Ultrasonic Bone Scalpel for Unilateral Cervical Open-Door Laminoplasty: A Randomized Controlled Trial. Neurosurgery. 2020 Jun 1;86(6):825-834. doi: 10.1093/neuros/nyz301. PMID 31435653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasonic Osteotome | Drill
Started | 95 | 95
Completed | 95 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients underwent cervical laminoplasty
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasonic Osteotome | Drill | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 58 (12) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 62 | 61 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 95 | 95 | 190
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 95 | 95 | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bone Fusion
Description: Bone fusion based on computed tomography scan taken at postoperative 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonic Osteotome | Drill
Number analyzed (Participants) | 95 | 95
Participants | 43 | 60

2. Secondary Outcome: Bleeding Amount
Description: bleeding amount through suction and gauze, unit mL
Time Frame: during operation
Population: bleeding amount through suction and gauze Date from all participants in this study
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Ultrasonic Osteotome: making gutter on the hinge side of lamina with ultrasonic osteotome
  ultrasonic osteotome: making gutter with ultrasonic osteotome
  mean 159.6 ml
- Drill: making gutter on the hinge side of lamina with conventional drill
  drill: making gutter with drill
  mean 139 ml
Arm/Group | Ultrasonic Osteotome | Drill
Number analyzed (Participants) | 95 | 95
ml | 159.6 (155.9) | 227.4 (139.5)

3. Secondary Outcome: Fracture of Laminar
Description: The number of patients with lamina fractures.
Time Frame: during operation
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonic Osteotome | Drill
Number analyzed (Participants) | 95 | 95
Participants | 23 | 25

4. Secondary Outcome: Neck Pain/Arm Pain
Description: Neck pain and arm pain were measured using a visual analogue scale (VAS), which is an integer with a minimum value of 0 and a maximum value of 10. Higher scores indicate a worse outcome.
Time Frame: postop 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasonic Osteotome | Drill
Number analyzed (Participants) | 78 | 75
score on a scale
  Neck pain | 2.15 (0.25) | 1.96 (0.25)
  Arm pain | 3.02 (0.29) | 2.39 (0.30)

5. Secondary Outcome: Functional Outcome
Description: Functional outcomes were assessed using the Neck Disability Index (NDI).
  The NDI consists of the following 10 subscales, each scored on a scale from 0 to 5:
  Pain intensity (range: 0-5) Personal care (range: 0-5) Lifting (range: 0-5) Reading (range: 0-5) Headaches (range: 0-5) Concentration (range: 0-5) Work (range: 0-5) Driving (range: 0-5) Sleeping (range: 0-5) Recreation (range: 0-5) Each subscale has a minimum score of 0 and a maximum score of 5, with higher values indicating worse outcomes.
  The total NDI score is calculated as the sum of all 10 subscale scores, ranging from 0 to 50. This total score is then converted into a percentage score (0-100%) by dividing the total score by 50 and multiplying by 100. Higher percentage scores indicate worse functional outcomes.
Time Frame: postop 1 year
Measure: Mean (Standard Deviation); unit: percentage score on a 0-100% scale
Arm/Group | Ultrasonic Osteotome | Drill
Number analyzed (Participants) | 78 | 75
percentage score on a 0-100% scale | 11.30 (0.95) | 10.79 (0.97)

ADVERSE EVENTS:
Time Frame: 1 year
Description: neurological deterioration, any unexpected complicaitons All those complication did not occur during follow-up period
Arm/Group | Ultrasonic Osteotome | Drill
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 0/95 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02487901/Prot_SAP_000.pdf